CLINICAL TRIAL: NCT04380610
Title: Improving Scientific Rigor of Renal Clinical Endpoints for Sickle Cell Anemia
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jeffrey D. Lebensburger, DO, PI, University of Alabama at Birmingham
Other Study IDs: IRB-300005433; 1R01HL153386 (NIH)
Record Dates: First submitted 2020-05-05; First posted 2020-05-08 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Sickle Cell Disease; Renal Disease; Glomerular Disease
MeSH Terms: conditions — Anemia, Sickle Cell; Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Pediatric SCA: We will develop a novel eGFR equation in 200 pediatric participants
  Interventions: Diagnostic Test: iohexol GFR
- Adult SCA: We will develop a novel eGFR equation in 200 adult participants
  Interventions: Diagnostic Test: iohexol GFR

INTERVENTIONS:
Diagnostic Test: iohexol GFR — We will perform mGFR in 400 SCA patients

SUMMARY:
The investigators will attempt to develop a more accurate equation to estimate eGFR in pediatric and adult sickle cell patients

DETAILED DESCRIPTION:
200 pediatric and 200 adult SCA participants will undergo mGFR using iohexol at baseline and at one year. On the same day, participants will undergo clinical and laboratory variables important for developing an eGFR equation. From baseline data, the investigators will perform a training and validation cohort of biologically relevant predictor variables to develop a novel equation. Then the investigators will compare the novel SCA eGFR equation to the established eGFR equation. From one year data, the investigators will determine the longitudinal concordance between pediatric and adult novel and standard eGFR equations with mGFR and variables that may alter longitudinal inferences.

In a subset of 30 adult participants, the investigators will also evaluate the correlation between mGFR using iohexol and a novel measure of mGFR that is more time efficient

ELIGIBILITY:
Inclusion Criteria:

* SCA patients (HbSS and SB0 thalassemia)
* Age: 5.0-50.0 at enrollment

Exclusion Criteria:

* Recent SCA complication associated with hospitalization (within 30 days) or ED visit (within 14 days)
* Current AKI defined as >0.3mg/g increase in SCr from prior visit
* Known history of anaphylaxis with contrast agent or known pregnancy

Ages: 5 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients with sickle cell anemia
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2021-05-12 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
To develop a novel SCA-specific eGFR equation and compare with existing eGFR equations validated for the general population | 5 years
  The investigators will use biologically relevant variables to develop a new equation for eGFR in pediatric and adult sickle cell patients

SECONDARY OUTCOMES:
To determine the longitudinal concordance between pediatric and adult novel and standard eGFR equations with mGFR and variables that may alter longitudinal inferences. | 5 years
  To compare the concordance between eGFR and mGFR from baseline to one year
To test the correlation of the novel mGFR method using VFI FAST and iohexol mGFR. | 5 years
  To perform a 3 hour mGFR and compare this mGFR to the 6 hour mGFR (iohexol)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Lebensburger, DO, MSPH, Principal Investigator — University of Alabama at Birmingham
Locations (4):
- United States (4):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Illinois Chicage, Chicago, Illinois
  - St Jude Childrens Research Hospital, Memphis, Tennessee
  - University of Tennessee Health Science Center, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Data collected in this study will be made available to other researchers, after the goals have been met and primary aims have been published. Disclosure of sensitive health and behavior data present a potential risk to human subjects, and we will take all steps to ensure that this does not happen when data are shared. In addition, we will strongly recommend that all recipient groups ensure that every member of the staff sign a Confidentiality Agreement. We will develop a data and resource sharing agreement with the legal advice from the Compliance Office of the UAB. Before data is shared with researchers, we will require that researchers enter into a data- and resource-sharing agreement. This agreement will ensure that: 1) data are used only for research purposes; 2) data do not identify any individual participant; 3) data are secure, using appropriate computer technology; and 4) there is a commitment to destroy or return data after analyses are completed.